CLINICAL TRIAL: NCT06580236
Title: Study of the Safety, Tolerability, Immunogenicity, Pharmacokinetics and Pharmacodynamics of the Drug B11-FC With a Single Application in Adults
Brief Title: Study of the Drug B11-FC (Botulism Treatment)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: № 01- B11-FC -2024
Record Dates: First submitted 2024-08-15; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-07

CONDITIONS: Botulism
MeSH Terms: conditions — Botulism | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Arm 1 - doze 1 (Experimental): B11-FC 0,06 mg/kg single infusion - 5 subjects
  Interventions: Drug: B11-FC
- Arm 2 - doze 2 (Experimental): B11-FC 0,3 mg/kg single infusion - 5 subjects
  Interventions: Drug: B11-FC
- Arm 3 - doze 3 (Experimental): B11-FC 0,6 mg/kg single infusion - 5 subjects
  Interventions: Drug: B11-FC
- Arm 4 - selected doze (Active Comparator): B11-FC 0,6 mg/kg single infusion + botulinum neurotoxin - 5 subjects
  Interventions: Drug: B11-FC; Drug: Botulinum neurotoxin type A
- Arm 5 - placebo (Placebo Comparator): Placebo + botulinum neurotoxin - 5 subjects
  Interventions: Drug: Botulinum neurotoxin type A; Other: Placebo
- Arm 6 - selected doze - patients with confirmed botulism (Active Comparator): B11-FC 0,6 mg/kg single infusion - 10 subjects
  Interventions: Drug: B11-FC

INTERVENTIONS:
Drug: B11-FC — Infusion
  Arms: Arm 1 - doze 1; Arm 2 - doze 2; Arm 3 - doze 3; Arm 4 - selected doze; Arm 6 - selected doze - patients with confirmed botulism
Drug: Botulinum neurotoxin type A — Infusion
  Arms: Arm 4 - selected doze; Arm 5 - placebo
Other: Placebo — Infusion
  Arms: Arm 5 - placebo

SUMMARY:
Study of the safety, tolerability, immunogenicity, pharmacokinetics and pharmacodynamics of the drug B11-FC with a single application in adults

DETAILED DESCRIPTION:
A three-staged, open-label, prospective study of B11-FC to examine safety, tolerability, immunogenicity, and pharmacokinetics in three dose-escalation groups; pharmacodynamics with a single dose in adult volunteers in a model of the effect of botulinum antitoxin on paralysis caused by botulinum neurotoxin A in EDB muscles in the framework of a double-blind, placebo-controlled comparative study and studying the effect of the study drug on the course of disease caused by botulinum toxin type A in adult patients diagnosed botulism.

The study plans to examine the safety of the drug after a single dose. The therapeutic dose is calculated based on the activity of monoclonal antibodies included in the drug. To ensure the safety of volunteers, drug administration will be started with 1/10 of the therapeutic dose.

The study for each participant of stages 1 and 2 consists of 3 periods:

* screening (no more than 7 days before drug administration);
* period of administration of the study drug and observation in a hospital setting (hospitalization for 7 days);
* follow-up period (from 8 to 90 days from the date of administration). A total of 9 visits will take place, including a screening visit, of which 1 visit will be carried out as part of inpatient observation, and 7 visits will be outpatient. During the visits, volunteers will be examined in accordance with the study plan.

The study design will be the same for all volunteers, with the exception of the dosing regimen.

The study for each participant of stage 3 consists of 3 periods:

* screening (on the day of hospitalization);
* period of administration of the study drug and observation in a hospital setting (hospitalization for at least 7 days);
* follow-up period (from the moment of discharge from the hospital to 90 days from the moment of administration).

During the visits, patients will be assessed and treated according to the study design and botulism treatment standards.

ELIGIBILITY:
Inclusion Criteria:

Volunteers who meet all the specified criteria will be included in the study of stages 1 and 2:

1. Healthy volunteers of both sexes aged 18 to 45 years (inclusive);
2. Provided signed Informed Consent prior to the initiation of any screening procedures, and the ability, in the opinion of the Investigator, to comply with all study requirements;
3. Body mass index (BMI) 18.5 - 29.9 kg/m2 inclusive;
4. Healthy according to the results of a medical examination: no history, as well as according to a screening examination, of pathologies of the gastrointestinal tract, liver, kidneys, cardiovascular system, central nervous system, musculoskeletal system, genitourinary, immune and endocrine systems, blood, which may affect the safety of the volunteer and the evaluation of the study results (clinical, instrumental and laboratory studies did not reveal diseases or deviations from reference values, including: hemodynamic parameters within normal limits: systolic blood pressure (BP) within 100-130 mmHg, diastolic blood pressure within 60-90 mmHg, heart rate - 60-90 beats/min, respiratory rate - 14-20 per minute, body temperature - 35.9-36.9°C; no deviations from the norm in the results of laboratory and instrumental examinations, including ECG).
5. Consent to use effective methods of contraception during the entire period of participation in the study (dual barrier method: male or female condom and combined hormonal contraceptive (oral, vaginal and transdermal forms can be used), or use of a condom or diaphragm with spermicide throughout the study period).
6. Negative pregnancy test based on urine test results at the screening visit (for women of reproductive age)
7. Negative tests for HIV, hepatitis B and C, syphilis;
8. Negative test for the presence of narcotic and psychostimulant drugs in the urine;
9. Negative alcohol test;
10. Indicators of general and biochemical blood tests during screening are within the range of 1.1 X VGRI - 0.9 X NGRI,
11. Immunoglobulin E levels are not higher than 2 X VGRI

    The Stage 3 study will include patients who meet all of the following criteria:
12. Patients of both sexes over 18 years old
13. Provided signed Informed Consent prior to the initiation of any screening procedures, and the ability, in the opinion of the Investigator, to comply with all study requirements;
14. Diagnosis of botulism

Exclusion Criteria:

Volunteers cannot be included in the Phase 1 study if at least one of the following non-inclusion criteria is met:

1. Inability to read Russian; inability or unwillingness to understand the essence of the study. Any other condition that limits the eligibility of obtaining informed consent or may affect the volunteer's ability to participate in the study;
2. History of botulism, repeated administration of high doses of botulinum neurotoxin type A for cosmetic or therapeutic purposes
3. Acute infectious diseases within 2 weeks and non-infectious diseases, exacerbations of chronic diseases within 4 weeks preceding screening;
4. The presence of changes in the myocardium of an inflammatory or dystrophic nature according to the results of an ECG during screening;
5. Volunteer participation in any other clinical trial within the last 90 days;
6. History of splenectomy.
7. Presence of mental illness (registered with a psychiatrist).
8. Treatment with steroids (excluding hormonal contraceptives) in the last 10 days;
9. Administration of monoclonal antibodies, immunoglobulins or blood products in the last 3 months;
10. History of autoimmune diseases or systemic collagenosis requiring immunosuppressive therapy.
11. Volunteers who have undergone an organ transplant, including bone marrow or peripheral blood stem cell (PBSC) transplantation.
12. Taking immunosuppressive drugs and/or immunomodulators within 6 months before the start of the study;
13. Any immunodeficiency (for example, hereditary immunodeficiency, acquired immunodeficiency syndrome [AIDS], etc.)
14. Systolic blood pressure less than 100 mmHg or above 130 mmHg; diastolic blood pressure less than 60 mmHg or above 90 mmHg; heart rate less than 60 beats/min or more than 90 beats/min;
15. Aggravated allergic history (history of anaphylactic shock, angioedema and other life-threatening conditions), hypersensitivity or allergic reactions to the administration of immunobiological drugs, exacerbation of allergic diseases on the day of inclusion in the study;
16. History of severe infusion reactions
17. Diabetes mellitus or other forms of impaired glucose tolerance;
18. Previously diagnosed or currently suspected multiple sclerosis or other neuromuscular degenerative disease
19. Previously diagnosed or currently suspected coagulopathies
20. Previously diagnosed or currently suspected vasculitis
21. A history of malignant neoplasms, with the exception of basal cell or squamous cell epithelial carcinomas of the skin, which were removed without signs of metastasis within 3 years;
22. Blood donation (450 ml or more of blood or plasma) less than 2 months before the start of the study;
23. Taking narcotic and psychostimulant drugs currently or in history;
24. Alcohol consumption exceeding the low-risk level: no more than 20 grams of pure alcohol per day, no more than 5 days a week, drinking alcohol within 48 hours before administration of the study drug;
25. Smoking: more than 10 cigarettes per day;
26. Planned hospitalization and/or surgical intervention during the period of participation in the study, as well as 4 weeks before the expected date of drug administration.
27. The presence of a concomitant disease that may affect the assessment of the study results or which, in the opinion of the investigator, will not allow the volunteer to participate in the study or may affect the conduct of the study and/or its results (including the assessment of safety parameters), any conditions that, in the opinion of the investigator's physician, may be a contraindication to participation in the study;
28. The volunteer's weight is less than 45 and more than 100 kg (even if the volunteer's BMI corresponds to the norm - clause 8 of the inclusion criteria).

    Additional criteria for non-inclusion in stage 2
29. Previously diagnosed or currently suspected motor neuron disease, peripheral neuropathy of the nerves of the lower extremities
30. Current skin infection/skin problems at the injection site (foot)
31. Scar tissue or tattooed skin over the extensor digitorum brevis muscles.
32. Abnormal (based on the principal judgment of the investigator) results of a nerve conduction study (NCS)
33. Any medical condition that may place the participant at risk of exposure to BoNT, including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other disease that may affect neuromuscular function
34. Previous treatment with botulinum toxin (BoNT) (any serotype) within the last 6 months
35. Known hypersensitivity to any of the components of the drug botulinum neurotoxin type A
36. Use of agents that may affect neuromuscular transmission, including calcium channel blockers, penicillamine, aminoglycosides, lincosamides, polymyxins, magnesium sulfate, anticholinesterases, succinylcholine and quinidine.

Volunteers cannot be included in the Stage 3 study if at least one of the following non-inclusion criteria is met:

1. Limitation of the legality of obtaining informed consent to participate in the study.
2. Duration of illness more than 7 days
3. Age under 18 years
4. Pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
heart rate | through study completion, an average of 1 year
  heart rate measurement
respiratory rate | through study completion, an average of 1 year
  respiratory rate measurement
blood pressure (both systolic and diastolic) | through study completion, an average of 1 year
  blood pressure measurement
ECG Cardiac rate (beats per minute) | through study completion, an average of 1 year
  ECG Cardiac rate (beats per minute) measurement
ECG RR Interval (ms) | through study completion, an average of 1 year
  ECG RR Interval (ms) measurement
ECG PQ interval (ms) | through study completion, an average of 1 year
  ECG PQ interval (ms) measurement
ECG QRS interval (ms) | through study completion, an average of 1 year
  ECG QRS interval (ms) measurement
ECG QT interval (ms) | through study completion, an average of 1 year
  ECG QT interval (ms) measurement

IPD SHARING:
Plan to Share IPD: No